CLINICAL TRIAL: NCT07174349
Title: The Use of an Uroselective Alpha-1-antagonist to Reduce the Incidence and Duration of Postoperative Urinary Retention Following Spine Surgery
Brief Title: Uroselective Alpha-1-Antagonist to Reduce the Incidence and Duration of Postoperative Urinary Retention Following Spine Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michelle J. Clarke, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-005742
Record Dates: First submitted 2025-09-12; First posted 2025-09-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Urinary Retention Postoperative
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Neurosurgical patients undergoing decompressive laminectomy and/or spinal fusion who will receive uroselective alpha-1-adrenergic receptor antagonist Tamsulosin
  Interventions: Drug: Uroselective alpha-1-adrenergic receptor antagonist
- Control Group (Placebo Comparator): Neurosurgical patients undergoing decompressive laminectomy and/or spinal fusion who will receive a placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Uroselective alpha-1-adrenergic receptor antagonist — Subjects will receive Tamsulosin (0.4 mg daily) beginning 5 days prior to surgery and for the duration of the postoperative hospital stay (approximately 8-12 days)
  Other Names: Tamsulosin
  Arms: Treatment Group
Other: Placebo — Subjects will receive placebo beginning 5 days prior to surgery and for the duration of the postoperative hospital stay (approximately 8-12 days)
  Arms: Control Group

SUMMARY:
The purpose of this research is to see if the use of tamsulosin can decrease both the incidence and duration of urinary retention, as well as hospital length of stay following spine surgery.

DETAILED DESCRIPTION:
Postoperative urinary retention is a frequent complication of spinal surgeries and impacts a large portion of this population which results in increased morbidity as a result of increased number of catheterizations, urinary tract infections and prolonged hospital stays. With the addition of Tamsulosin, we would anticipate a reduction in the incidence and duration of postoperative urinary retention and therefore a reduction in morbidity related to treatment of urinary retention as well as shortened hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Laminectomy
* Cervical Posterior Fusion
* Cervical Anterior/Posterior Fusion
* Lumbar Laminectomy
* Lumbar Posterolateral Fusion
* Lumbar Interbody Fusion

Exclusion Criteria:

* Cervical Anterior Discectomy and Fusion
* Cervical Anterior Corpectomy
* Cervical Posterior Discectomy
* Cervical Foraminotomy
* Lumbar Discectomy (METRx or Open)
* Lumbar Foraminotomy
* Lumbar Anterior Fusion
* Myelopathy with bladder dysfunction
* Patients currently taking an alpha-antagonist

  o The following drugs are alpha antagonists: alfuzosin, doxazosin, prazosin, terazosin, tamsulosin, and phenoxybenzamine.
* Patients with history of allergy or sensitivity to tamsulosin or other alpha-antagonist
* History of prostatectomy or urologic surgery involving the bladder or urethra
* Severe liver disease or end-stage renal disease
* Patients taking strong inhibitors of CYP3A4

  o The following drugs are strong inhibitors of CYP3A4: ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir/ritonavir, lopinavir/ritonavir, and conivaptan.
* Mental disability or prisoner
* Pregnancy (for anesthesia purposes)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of incidences of POUR (Postoperative urinary retention) | Post-operatively through end of hospital stay, approximately 8-12 days
  Total number of incidences of POUR (Postoperative urinary retention). POUR is defined as any of the following: estimated post-void residual (PVR) volume of urine greater than or equal to 300 mL; estimated retention urine volume of greater than or equal to 500 mL in patients unable to void; or patients experiencing discomfort or distension and unable to void with lesser residual urine volume than 500 ml.

SECONDARY OUTCOMES:
Duration of POUR (Postoperative urinary retention) | Post-operatively through end of hospital stay, approximately 8-12 days
  Duration subjects experience postoperative urinary retention, reported in days
Number of intermittent catheterizations in those with urinary retention | Post-operatively through end of hospital stay, approximately 8-12 days
  Total number of catheterizations performed in subjects who experience urinary retention
Incidence of UTI (urinary tract infection) | Post-operatively through end of hospital stay, approximately 8-12 days
  Number of subjects to be diagnosed with a UTI (urinary tract infection) post-operatively
Duration of hospital stay | Post-operatively through end of hospital stay, approximately 8-12 days
  Total length of time subjects remain inpatient post-procedure, reported in days.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Clarke, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials